CLINICAL TRIAL: NCT01500252
Title: A Randomized Clinical Trial Comparing Patellar Resurfacing Versus Patellar Retention in Total Knee Arthroplasty Using the PROFIX* Total Knee System
Brief Title: Patellar Resurfacing Versus Patellar Retention in Total Knee Arthroplasty - A Randomized Clinical Trial
Acronym: PROFIX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00002794
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Total Knee Replacement
Keywords: Total Knee Replacement; Patellar Resurfacing; Health Related Quality of Life

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patellar Resurfacing (Experimental): These subjects received a Profix TKR including an all polyethylene patellar implant.
  Interventions: Device: Patellar Replacement Prosthesis
- Patellar Retention (Active Comparator): This group received a Profix TKR, but retained their native patella
  Interventions: Device: Profix TKR with Patellar Retention

INTERVENTIONS:
Device: Patellar Replacement Prosthesis — The Profix™ Total Knee System, a posterior cruciate retaining prosthesis manufactured by Smith and Nephew, Inc. was utilized in all subjects. Subjects randomized to the Resurfaced group received an all polyethylene patellar implant
  Arms: Patellar Resurfacing
Device: Profix TKR with Patellar Retention — All subjects received a Profix TKR. Subjects in the Patellar Retention group retained their native patellar surface.
  Arms: Patellar Retention

SUMMARY:
Background:

Despite the excellent results of total knee replacement, also known as total knee arthroplasty (TKA) there is persistent controversy over whether or not to replace the surface of the kneecap. Anterior knee pain, which occurs with variable and unpredictable frequency, continues to be a problem in a subset of TKA patients. Some clinicians replace the surface of all kneecaps during TKA to avoid repeat surgery, which occurs in approximately 10% of cases. However, others cite the complications attributed to replacing the surface of kneecap as reasons to avoid this procedure.

This study prospectively randomized patients receiving TKA into two groups, those receiving replacement of the kneecap surface and those left without replacement of the kneecap surface to determine clinical outcomes and revisions over the first 5-10 postoperative years.

Objectives:

The primary objective of this work was to compare pain, stiffness and function between groups at five years postoperatively. Secondarily, we compared pain, stiffness and function at one and 10 years postoperatively. Finally, we examined the number of reoperations following TKR over 10 years in the 2 groups of subjects. The investigators hypothesized that there would be no difference between the two groups of subjects in the measured outcomes.

Methods:

Patients receiving TKA were prospectively enrolled before surgery and randomized intraoperatively to either receive a replacement of the kneecap surface or have no kneecap intervention. The Smith and Nephew Profix TKA system was implanted in all cases; the post-operative regimen was standardized. Subjects were assessed pre-operatively and at 1 and 5 years postoperatively for pain, function, and stiffness using a disease-specific (Western Ontario and MacMaster Osteoarthritis Index [WOMAC]) and generic health status (Short Form 36 [SF-36]) questionnaire. At the end of the five year follow-up, the study was extended to a 10-year followup and the same outcomes were assessed. The revision rate was also compared between the two groups at the end of the 10-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for primary TKA to treat non-inflammatory arthritis
* age 40- 75 years of age

Exclusion Criteria:

* history of knee sepsis
* previous patellectomy
* previous high tibial osteotomy
* knee flexion contracture of >20 degrees
* varus or valgus deformity of > 20 degrees
* < 90 degrees of knee flexion
* tibial or femoral bone deficiency requiring augmentation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1996-09; Primary Completion 2004-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Beaupre L, Secretan C, Johnston DW, Lavoie G. A randomized controlled trial comparing patellar retention versus patellar resurfacing in primary total knee arthroplasty: 5-10 year follow-up. BMC Res Notes. 2012 Jun 7;5:273. doi: 10.1186/1756-0500-5-273. PMID 22676495

RESULTS

PARTICIPANT FLOW:
Groups:
- Patellar Resurfacing: Subjects received patellar resurfacing.
- Patellar Retention: Subjects retained their native patella.
Period: Overall Study
Arm/Group | Patellar Resurfacing | Patellar Retention
Started | 21 | 17
One Years | 20 | 16
Five Years | 17 | 13
Ten Years | 12 | 11
Completed | 12 (2 participants died within 5 years; 2 participants died between 5 & 10 years for a total of 4 deaths) | 11 (2 participant deceased by 5 years; no further deaths between 5 & 10 years for a total of 2 deaths)
Not Completed | 9 | 6
Not completed — Death | 4 | 2
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patellar Resurfacing | Patellar Retention | Total
Number analyzed (Participants) | 21 | 17 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 13 | 22
  >=65 years | 12 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (4.0) | 62.0 (5.6) | 63.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Western Ontario MacMaster (WOMAC) Osteoarthritis Index Pain Score From Preoperative to 5 Years Postoperative
Description: This index assesses pain as reported by the patient. The WOMAC Pain scale has a minimum value of 0 (worst pain) to a maximum value of 100 (no pain).
  The change score was calculated by subtracting the preoperative score from the five year score.
Time Frame: Preoperative to 5 years postoperative
Population: One subject in the patellar retention group missed too many responses on the WOMAC questionnaire and was not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 17 | 12
units on a scale | 34.7 (20.9) | 39.2 (19.6)
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.59, t-test, 2 sided

2. Secondary Outcome: Change in WOMAC Osteoarthritis Index Pain Score From Preoperative to 1 Year Postoperative
Description: This index assesses pain as reported by the patient. The WOMAC Pain scale has a minimum value of 0 (worst pain) to a maximum value of 100 (no pain).
  The change score was calculated by subtracting the preoperative score from the one year score.
Time Frame: Preoperative to 1 year postoperative
Population: Two subjects, one in the patellar retention group and one in the patellar resurfacing group missed too many responses on the WOMAC questionnaire and was not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 19 | 15
units on a scale | 32.9 (18.2) | 34.3 (21.5)
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.83, t-test, 2 sided

3. Secondary Outcome: Change in WOMAC Osteoarthritis Index Function Score From Preoperative to 1-year Postoperative
Description: This index assesses function as reported by the patient. The WOMAC function scale has a minimum value of 0 (worst function) to a maximum value of 100 (no functional limitations).
  The change score was calculated by subtracting the preoperative score from the one year score.
Time Frame: Preoperative to 1 year postoperative
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 19 | 15
units on a scale | 24.1 (16.6) | 19.5 (16.9)

4. Secondary Outcome: Change in WOMAC Osteoarthritis Index Stiffness Score From Preoperative to 1 Year Postoperative
Description: This index assesses stiffness as reported by the patient. The WOMAC stiffness scale has a minimum value of 0 (worst stiffness) to a maximum value of 100 (no stiffness).
  The change score was calculated by subtracting the preoperative score from the one year score.
Time Frame: Preoperative to 1 year postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 19 | 15
units on a scale | 24.4 (24.5) | 8.3 (32.3)
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.10, t-test, 2 sided

5. Primary Outcome: Change in WOMAC Osteoarthritis Index Function Score From Preoperative to 5 Years Postoperative
Description: This measures the change in patients' reported function from preoperative to 5 years postoperative.
  The WOMAC Function scale has a minimum value of 0 (worst function) to a maximum value of 100 (no functional limitations).
  The change score was calculated by subtracting the preoperative score from the five year score.
Time Frame: Preoperative to 5 years postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 17 | 12
units on a scale | 21.8 (17.9) | 27.5 (15.6)
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.39, t-test, 2 sided

6. Primary Outcome: Change in WOMAC Osteoarthritis Index Stiffness Score From Preoperative to 5 Years Postoperative
Description: This is the change in the patients' perceived pain between preoperative and 5 years postoperative.
  The WOMAC stiffness scale has a minimum value of 0 (maximal stiffness) to a maximum value of 100 (no stiffness).
  The change score was calculated by subtracting the preoperative score from the five year score.
Time Frame: Preoperative to 5 years postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 17 | 12
units on a scale | 38.2 (32.0) | 29.2 (26.3)
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.43, t-test, 2 sided

7. Secondary Outcome: Change in WOMAC Osteoarthritis Index Pain Score From 5 Years Postoperative to 10 Years Postoperative
Description: This index assesses pain as reported by the patient. The WOMAC Pain scale has a minimum value of 0 (worst pain) to a maximum value of 100 (no pain).
  The change score was calculated by subtracting the five year score from the 10 year score.
Time Frame: 5 years postoperative to 10 years postoperative
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 12 | 11
units on a scale | 12.7 (20.0) | 10.0 (12.0)
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.71, t-test, 2 sided

8. Secondary Outcome: Change in WOMAC Osteoarthritis Index Function Score From 5 Years Postoperative to 10 Years Postoperative
Description: This index assesses function as reported by the patient. The WOMAC function scale has a minimum value of 0 (worst pain) to a maximum value of 100 (no pain).
  The change score was calculated by subtracting the five year score from the 10 year score.
Time Frame: 5 years postoperative to 10 years postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 12 | 11
units on a scale | 14.2 (17.7) | 14.4 (13.6)
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.98, t-test, 2 sided

9. Secondary Outcome: Change in WOMAC Osteoarthritis Index Stiffness Score From 5 Years Postoperative to 10 Years Postoperative
Description: This index assesses stiffness as reported by the patient. The WOMAC stiffness scale has a minimum value of 0 (worst stiffness) to a maximum value of 100 (no stiffness).
  The change score was calculated by subtracting the five-year score from the 10 year score.
Time Frame: 5 years postoperative to 10 years postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 12 | 11
units on a scale | 3.4 (33.6) | 15.0 (19.4)
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.35, t-test, 2 sided

10. Secondary Outcome: Number of Revision Surgeries
Description: This measure examined the number of reoperation in the two groups of subjects
Time Frame: 10 years
Population: All participants were analyzed.
Measure: Number; unit: participants
Arm/Group | Patellar Resurfacing | Patellar Retention
Number analyzed (Participants) | 21 | 17
participants | 3 | 1
Statistical Analysis 1: Comparison: Patellar Resurfacing vs Patellar Retention; Test type: Superiority or Other; p = 0.31, Chi-squared

ADVERSE EVENTS:
Arm/Group | Patellar Resurfacing | Patellar Retention
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/17
Other Adverse Events (participants affected / at risk) | 0/21 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No